CLINICAL TRIAL: NCT00057135
Title: Improving Antipsychotic Adherence Among Patients With Schizophrenia
Brief Title: Improving Antipsychotic Adherence Among Patients With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIR 01-074
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: Schizophrenia; Treatment Refusal; Drug Packaging; Reminder Systems; Antipsychotic Agents
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Treatment Refusal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Unit of use medication packaging; Behavioral: Mailed reminders to patient when medication refills are due; Behavioral: Note to Mental Health Provider when refill is overdue; Procedure: Aligning all prescriptions to fall due on same date

INTERVENTIONS:
Behavioral: Unit of use medication packaging
Behavioral: Mailed reminders to patient when medication refills are due
Behavioral: Note to Mental Health Provider when refill is overdue
Procedure: Aligning all prescriptions to fall due on same date

SUMMARY:
This is a randomized controlled trial examining the effectiveness of a pharmacy-based intervention designed to improve adherence with antipsychotic medications among patients with serious mental illness.

DETAILED DESCRIPTION:
Background: Anti-psychotic medications are an essential component of the treatment of patients with schizophrenia. Unfortunately, pharmacy data indicate that 40% of VA patients with schizophrenia are poorly adherent with their antipsychotics. These patients are at much greater risk for hospitalization. Objectives: We are examining the effectiveness of a practical, pharmacy-based intervention for improving antipsychotic adherence among patients with serious mental illness (SMI). Specifically, we are examining whether this pharmacy-based intervention increases antipsychotic medication adherence and patient satisfaction with care and decreases psychiatric symptoms, and inpatient utilization. We are also examining the relative effectiveness of the pharmacy-based intervention among patients with varying: a) degrees of cognitive limitations, b) degrees of insight into their illness, and c) attitudes towards their medications. Methods: Using pharmacy and administrative data, we are identifying patients with schizophrenia, schizoaffective disorder, or severe bipolar disorder requiring antipsychotic medication who have had poor antipsychotic adherence in the previous year. Patients must have completed at least two outpatient psychiatric visits at one of the study sites. Patients are randomized to: 1) usual care; or 2) the Pharmacy Based intervention. The pharmacy-based intervention consists of usual care plus: 1) "unit-of-use" adherence packaging; 2) a patient education session; 3) refill reminders; and 4) clinician notification of missed fills. In-person patient assessments are conducted at baseline, 6 months, and 12 months following randomization. Medical record and administrative data will be collected at baseline, 6 months, 12 months, and 18 months following randomization. The primary outcome measure is medication adherence as measured by the medication possession ratio and adherence categories which combine pharmacy information with patient self-report and antipsychotic blood levels. Patients� level of psychiatric symptoms, quality of life, and satisfaction are secondary outcome measures. In supplemental analyses, we will compare the effectiveness of the pharmacy-based intervention among subgroups of patients who have varying degrees of cognitive limitations, insight into their illness, and attitudes towards antipsychotic medication. Findings: One hundred and fifty patients have been enrolled in the study. Follow-up rates have been high, with 90% of patients completing 6 month follow up assessments and 80% completing 12 month assessments. In person follow up visits are now complete.

Findings regarding the accuracy of administrative diagnoses of schizophrenia, the accuracy of pharmacy data in identifying patients with poor adherence, and patient factors associated with study recruitment have been presented at national meetings. Main study analyses are now ongoing. 6. Status: Enrollment and inperson-patient follow up are complete. Study analyses are now in progress. Impact: Improving adherence among SMI patients is critical to improving their outcomes. This study examines the effectiveness of a practical, low-cost intervention to for these vulnerable patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must be adult veterans. Diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder. At least one active oral antipsychotic prescription. History of poor medication compliance.

Exclusion Criteria:

Have received depot antipsychotics in the last year. Have supervised medication administration. Have not attended a VA outpatient appointment in the past 6 months, and none are scheduled,. Are prescribed Clozapine. Have a fatal illness with a life expectancy less than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2002-11; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Medication Possession Ratio at baseline, 1-6 months, 6-12 months, and 12-18 months. Aggregate adherence categories based on MPR, anti-psychotic blood levels (present/not present) and patient self-report at baseline, 6 months, and 12 months.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale for Schizophrenia, Client Satisfaction Questionnaire, Quality of Well-Being Scale. All to be administered at baseline, 6 months, and 12 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Marcia T. Valenstein, MD AB, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; John Grabowski, MD, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (5):
- United States (5):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Rhode Island

REFERENCES:
- [Result] Kreyenbuhl J, Valenstein M, McCarthy JF, Ganoczy D, Blow FC. Long-term combination antipsychotic treatment in VA patients with schizophrenia. Schizophr Res. 2006 May;84(1):90-9. doi: 10.1016/j.schres.2006.02.023. Epub 2006 May 2. PMID 16631354
- [Result] Milner KK, Valenstein M. A comparison of guidelines for the treatment of schizophrenia. Psychiatr Serv. 2002 Jul;53(7):888-90. doi: 10.1176/appi.ps.53.7.888. PMID 12096176
- [Result] Sajatovic M, Valenstein M, Blow FC, Ganoczy D, Ignacio RV. Treatment adherence with antipsychotic medications in bipolar disorder. Bipolar Disord. 2006 Jun;8(3):232-41. doi: 10.1111/j.1399-5618.2006.00314.x. PMID 16696824
- [Result] Sajatovic M, Blow FC, Kales HC, Valenstein M, Ganoczy D, Ignacio RV. Age comparison of treatment adherence with antipsychotic medications among individuals with bipolar disorder. Int J Geriatr Psychiatry. 2007 Oct;22(10):992-8. doi: 10.1002/gps.1777. PMID 17323327
- [Result] Kreyenbuhl JA, Valenstein M, McCarthy JF, Ganoczy D, Blow FC. Long-term antipsychotic polypharmacy in the VA health system: patient characteristics and treatment patterns. Psychiatr Serv. 2007 Apr;58(4):489-95. doi: 10.1176/ps.2007.58.4.489. PMID 17412850
- [Result] Valenstein M, Ganoczy D, McCarthy JF, Myra Kim H, Lee TA, Blow FC. Antipsychotic adherence over time among patients receiving treatment for schizophrenia: a retrospective review. J Clin Psychiatry. 2006 Oct;67(10):1542-50. doi: 10.4088/jcp.v67n1008. PMID 17107245
- [Result] Sajatovic M, Valenstein M, Blow F, Ganoczy D, Ignacio R. Treatment adherence with lithium and anticonvulsant medications among patients with bipolar disorder. Psychiatr Serv. 2007 Jun;58(6):855-63. doi: 10.1176/ps.2007.58.6.855. PMID 17535948
- [Result] Valenstein M, Kavanagh J, Lee T, Reilly P, Dalack GW, Grabowski J, Smelson D, Ronis DL, Ganoczy D, Woltmann E, Metreger T, Wolschon P, Jensen A, Poddig B, Blow FC. Using a pharmacy-based intervention to improve antipsychotic adherence among patients with serious mental illness. Schizophr Bull. 2011 Jul;37(4):727-36. doi: 10.1093/schbul/sbp121. Epub 2009 Nov 21. PMID 19933540
- [Result] Pfeiffer PN, Szymanski B, Dhawan N, Difranco D, Valenstein M, Zivin K. Is there an "unhealthy volunteer effect" in mental health outpatient research? Psychiatry Res. 2010 Apr 30;176(2-3):224-8. doi: 10.1016/j.psychres.2009.07.016. Epub 2010 Feb 1. PMID 20122743